CLINICAL TRIAL: NCT00854438
Title: Pharmacist-initiated Reduction of Anticholinergic Drug Activity
Brief Title: Reduction of Adverse Events of Anticholinergic Drugs by Multidisciplinary Medical Reviews in Norwegian Nursing Homes
Acronym: PRADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Directorate of Health (Other Government)
Responsible Party: Principal Investigator, Torgeir Bruun Wyller, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1110
Record Dates: First submitted 2009-02-23; First posted 2009-03-03 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Anticholinergic Side Effects
Keywords: anticholinergic drugs; adverse events; elderly; clinical pharmacist; Evaluate the clinical effects of reducing anticholinergic in elderly
MeSH Terms: interventions — Physicians

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment arm (Experimental): Reduction of anticholinergic drug effects by pharmacist review
  Interventions: Other: Multidisciplinary drug reviews by pharmacist and physician
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Multidisciplinary drug reviews by pharmacist and physician — Reduction of anticholinergic drug effects by pharmacist review
  Arms: Active treatment arm

SUMMARY:
Thesis: Is drug-induced anticholinergic activity additive resulting in a total anticholinergic load causing harmful side effects in old, fragile patients? Is it possible to reduce the anticholinergic load by multidisciplinary medical review including a pharmacist and a physician? The effects of the medical reviews are measured by cognitive tests (MMS and CERADS word lists), a measure of mouth dryness, serum levels of anticholinergic activity, activity of daily living and neuropsychiatric symptoms.

Design: A randomized, controlled, single blinded interventional study in Norwegian nursing homes.

DETAILED DESCRIPTION:
Several studies have claimed that drugs showing anticholinergic activity in vitro cause high levels of serum anticholinergic activity in vivo that might cause impaired cognitive and functional functions in elderly. Pathophysiological changes in Alzheimer's dementia makes these patients particularly vulnerable for anticholinergic cognitive impairments. The PRADA-study is the first interventional study evaluating the clinical effects of reducing drug-induced anticholinergic load in patients with dementia. This is also the first interventional study in the Nordic countries evaluating the clinical effects of clinical pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Long-term nursing home patients with none, mild or moderate dementia (evaluated by CDR9,using drugs with a total anticholinergic burden that might lead to adverse events.

Exclusion Criteria:

* Not able to perform the testes because of physical or psychiatric illnesses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
CERADS word list measuring immediately and delayed recall | 4 years

SECONDARY OUTCOMES:
Mouth dryness | 4 years
ADL | 4 years
Serum anticholinergic activity | 4 years
CERADS word list recognition | 4 years
MMSE | 4 years
NPI | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir B. Wyller, Professor, Study Director — Ullevaal University Hospital; Hege Kersten, MScPharm/PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway